CLINICAL TRIAL: NCT03721185
Title: Efficacy of a Lipolytic Cream in the Body Composition of an Overweight and Obesity Treatment
Brief Title: Efficacy of a Lipolytic Cream in an Overweight and Obesity Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BiomediKcal (Other)
Collaborators: University of Alicante (Other); Universidad Miguel Hernandez de Elche (Other); Universidad Simón Bolívar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCE24918
Record Dates: First submitted 2018-09-24; First posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Lipolysis; Overweight and Obesity; Diet Modification; Physical Activity
Keywords: obesity; overweight; fat percentage; body fat; lipolytic cream
MeSH Terms: conditions — Overweight; Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: open-label, randomized, parallel-group
Masking Description: Researchers assessed the efficacy of a lipolytic cream with hypocaloric diet and physical activity in the treatment of overweight and obesity. The control treatment was lypolitic cream with hypocaloric diet and physicial activity and hypocaloric diet and physicial activity alone. In total, 102 patients were recruited and allocated to treatment (51: lypolitic cream with hypocaloric diet and physicial activity and, 51: hypocaloric diet and physicial activity alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LC (Active Comparator): Lypolitic cream with hypocaloric diet and physicial activity in 51 patients
  Interventions: Combination Product: Dr.K. Treatment
- NLC (Placebo Comparator): Hypocaloric diet and physicial activity alone in 51 patients
  Interventions: Combination Product: Dr.K. Treatment

INTERVENTIONS:
Combination Product: Dr.K. Treatment — Overweight and obesity treatment response

SUMMARY:
The coadyouvant efficacy of a combination of cosmetics ingredients in the form of a lipolytic cream with hypocaloric diet and physical activity were assessed and compared with with hypocaloric diet and physical activity for overweight and obesity treatment in patients.

DETAILED DESCRIPTION:
The coadyouvant efficacy and safety of a combination of cosmetics ingredients in the form of a lipolytic cream with hypocaloric diet and physical activity were assessed and compared with with hypocaloric diet and physical activity for overweight and obesity treatment in patients of both gender and different age groups. DESIGN: In a monocenter, open-label, randomized, parallel-group study of 102 patients that consulted for overweight and obesity treatment were analyzed in perimeters and body composition for 12 consecutive weeks that were medically prescribed a weekly hypocaloric diet and physical activity for one group of 51 patients, and hypocaloric diet, physical activity and the lypolitic cream at least twice per day for the other group of 51 patients. Efficacy was evaluated by comparing intial and final of all values in both groups. Safety was monitored by the incidence of adverse events. Patients also assessed the acceptability of the cream presentation.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and obesity treatment voluntary assistance

Exclusion Criteria:

* Hearth disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2018-09-23 (Actual)

PRIMARY OUTCOMES:
Change in body composition with a scientific impedanciometer | Baseline and weeks: 1, 4, 8, 12,16
  Body fat in kilograms and percentage variation measured with an impendaciometer (Tanita MC780)

SECONDARY OUTCOMES:
Change in perimeters measured with measuring tape | Baseline and weeks: 1, 4, 8, 12,16
  Variation in the perimeters in centimeters in waist, hip, thigh and arm.

IPD SHARING:
Plan to Share IPD: Yes
Anonymous patient information will be shared only if requested and justified in writing by researchers. It will be evaluated in committee if it is a justified request.
Supporting Information: SAP, ICF

REFERENCES:
- [Result] Byun SY, Kwon SH, Heo SH, Shim JS, Du MH, Na JI. Efficacy of Slimming Cream Containing 3.5% Water-Soluble Caffeine and Xanthenes for the Treatment of Cellulite: Clinical Study and Literature Review. Ann Dermatol. 2015 Jun;27(3):243-9. doi: 10.5021/ad.2015.27.3.243. Epub 2015 May 29. PMID 26082579
- [Result] Escudier B, Fanchon C, Labrousse E, Pellae M. Benefit of a topical slimming cream in conjunction with dietary advice. Int J Cosmet Sci. 2011 Aug;33(4):334-7. doi: 10.1111/j.1468-2494.2010.00630.x. Epub 2011 Feb 1. PMID 21284660
- [Result] Salavert M, Amarger S, Le Bouedec MC, Roger H, Souteyrand P, D'incan M. Allergic contact dermatitis to guggul in a slimming cream. Contact Dermatitis. 2007 May;56(5):286-7. doi: 10.1111/j.0105-1873.2006.00885.x. No abstract available. PMID 17441853